CLINICAL TRIAL: NCT01248260
Title: Preventing Fetal Body and Brain Size Reduction in Low-income Smoking Mothers: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamisu Salihu (Other)
Responsible Party: Sponsor-Investigator, Hamisu Salihu, Principal Investigator, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1KG14
Record Dates: First submitted 2010-11-10; First posted 2010-11-25 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Fetal Body Size; Fetal Brain Size
Keywords: Fetal body size; Fetal brain size; Folic acid
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher-strength folic acid (Experimental): Higher-strength folic acid (4mg).
  Interventions: Dietary Supplement: Folic Acid
- Low-strength folic acid (No Intervention): Low-strength (0.8mg) folic acid (standard of care)

INTERVENTIONS:
Dietary Supplement: Folic Acid — 4mg of higher strength folic acid once a day until delivery
  Arms: Higher-strength folic acid

SUMMARY:
The purpose of this study is to find out if folic acid prevents of the reduction of fetal body and brain size in infants whose mothers smoke.

DETAILED DESCRIPTION:
Smoking during pregnancy remains a common practice despite smoking cessation programs offered to mothers. Only 20-40% of women quit smoking during pregnancy which implies that a majority of smokers continue smoking despite the associated feto-infant morbidity and mortality. It is therefore important to identify ways and means of protecting these infants as they grow and develop during intrauterine life. In this study, we propose to assess the utility of higher-strength folic acid (4mg) combined with smoking cessation programs as compared to standard of care (smoking cessation program and low-strength (0.8mg) folic acid) in reducing the level of morbidity (specifically fetal body and brain size) sustained by infants of smokers

ELIGIBILITY:
Inclusion Criteria:

((1) Smoker, based on presence of detectable cotinine in saliva (biomarker).; (2) Ages 18-44 years; (3) Singleton gestation (< 20 weeks), confirmed by sonogram; (4) Residents of Tampa, Florida or surrounding area in order to facilitate follow-up and reduce attrition rate.

Exclusion Criteria:

(a) an indication for chronic blood transfusion. Women receiving chronic blood transfusions will not be enrolled, as transfused red blood cells (RBC) can result in inaccurate analysis of folate RBC levels88; (b) generalized seizure disorder treated with anti-convulsant medication: Patients with generalized seizure disorder treated with anticonvulsant medication will be excluded because of the potential association with folic acid deficiency88.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 495 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Fetal Body Size | Participants will be followed from baseline (first trimester) until delivery
  Low birth weight will be defined as birth weight less than 2500g; Small for gestational age will be defined as birth weight in the lowest 10th percentile; The fetal growth ratio will be expressed as the ratio of the observed birth weight to the expected mean birth weight for each gestational age.
Fetal Brain Size | Participants will be followed from baseline (first trimester) until delivery
  Head Circumference at birth: will be measured at birth as routinely performed at the study site. Observed: Expected head circumference ratio: This is the ratio between the actual head circumference and the expected head circumference according to gestational age (this could also be expressed in terms of percentage of expected head circumference). Brain weight: will be estimated from formula: brain weight (g) = 0.037 X head circumference (cm)2.57. Brain-to-body ratio (BBR): The BBR is defined as 100 the ratio of the infant's estimated brain weight to its birth weight.

SECONDARY OUTCOMES:
Preterm Birth | Participants will be followed from baseline (first trimester) until delivery
  This is defined as live birth after 20 weeks of gestation but before 37 completed weeks. Genetic and Epigenetic Markers of Fetal Brain Growth and Development: Cord blood obtained at delivery will be analyzed for selected regulatory genes.

CONTACTS AND LOCATIONS:
Overall Officials: Hamisu M Salihu, MD, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, College of Public Health, Department of Epidemiology and Biostatistics, Tampa, Florida, United States

REFERENCES:
- [Derived] Yusuf KK, Salihu HM, Wilson R, Mbah A, Sappenfield W, Bruder K, Wudil UJ, Aliyu MH. Folic Acid Intake, Fetal Brain Growth, and Maternal Smoking in Pregnancy: A Randomized Controlled Trial. Curr Dev Nutr. 2019 Apr 4;3(6):nzz025. doi: 10.1093/cdn/nzz025. eCollection 2019 Jun. PMID 31139766